CLINICAL TRIAL: NCT05337501
Title: Prognostic Factors for Complex Regional Pain Syndrome: a Longitudinal Study
Brief Title: Prognostic Factors for Complex Regional Pain Syndrome
Acronym: CRPSPrognosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/28FEV/093
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective longitudinal observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients group (Experimental)
  Interventions: Other: Collecting data

INTERVENTIONS:
Other: Collecting data — Anamnesis, clinical examination, Quantitative Sensory Testing (following DFNS, German Research Network on Neuropathic Pain, protocol), visual TOJ (Temporal Order Judgement) task

SUMMARY:
The investigators would like to examine the role of some relevant biopsychosocial factors in the development of persistent CRPS. According to the International Classification of Functioning, Disability and Health (ICF) [43], the outcomes will belong to one of the three following components:

* Body structures and functions (pain, CRPS severity score (CSS)),
* Activities (disability)
* Participation (return to work, quality of life). The primary aim is to assess predicting factors for chronification.

The secondary aims are:

* to evaluate if it is possible to classify acute complex regional pain syndrome (CRPS) patients into subgroups according to their risk of chronification.
* to document the course of the disease. The main evaluation criteria will be to determine the impact of the different clinical and non-clinical variables on the course of the CRPS and on the aforementioned outcomes then, which will use as endpoints.
* Primary endpoint: disability
* Secondary endpoints: participation-QoL, return to work, pain, CRPS severity score.

DETAILED DESCRIPTION:
Patients suffering from early CRPS will be invited to attend 4 medical interviews over a 1-year period. A series of clinical data will be collected during this interview. After each consultation, the patient will be asked to complete a series of questionnaires at home (paper forms or online by REDCap). These questionnaires assess various psychosocial factors well known in the chronification of pain (fear of movement, anxious or depressive traits, "general" pain sensitization, social support, cognitive strategies to cope with pain) as well as the functional impact of the pathology.

All the study (first face-to-face assessment or follow-up sessions) will take place at Institute of Neurosciences (UCLouvain, site Woluwé) and perform by Pr. Berquin or Dr. Louis. As part of the study, the patients will never be assessed in another location or by another investigator.

After having encoded the patients' details in the REDCap application, the participants will receive an automatic e-mail at every time point. It will include a link to the online survey. At any given moment of the study, they can contact the co-investigator (Dr. Louis) by e-mail or phone for any questions or help in completing the questionnaires. If necessary, the co-investigator will provide assistance by telephone

To simplify the recruitment process, the informed consent will be sent by post or e-mail and signed during the first meeting.

Five endpoints will be tested using linear mixed-effects regression models for repeated measures:

Primary endpoint: disability Secondary endpoints: participation-QoL, return to work, pain, CRPS severity score.

A latent profiles analysis will be performed to classify patients into subgroups based on variables at baseline and the risk of chronicity of profile will be computed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18,
2. Meeting the clinical Budapest criteria,
3. Apparition of symptoms from less than 6 months,
4. CRPS type I or II,
5. Capacity to understand and voluntarily sign an informed consent form in French.

Exclusion Criteria:

1. Insufficient French language skills to answer questionnaires,
2. Personal history of CRPS at the same limb,
3. Post-stroke CRPS type I ("shoulder-hand syndrome"),
4. Psychiatric disorders that would interfere with the participants' ability to complete study tasks,
5. The following hormonal situations: gravidity, lactation, gender-affirming treatment,
6. Any other reason to exclude the subject because it may interfere with the study, according to judgment by the investigator. The reason will be documented.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Disability | 12 months
  Defined by International Classification of Functioning, Disability and Health (ICF), assessed by Quick DASH (0 to 100 scale) or Lower Extremity Functional Scale (LEFS) (0 to 80 scale) ; higher score means higher disability

SECONDARY OUTCOMES:
Participation - QoL | 12 months
  Defined by International Classification of Functioning, Disability and Health (ICF), assessed by EuroQol5D5L ; higher score in each domain means lower QoL ; lower score in visual analogic scale means lower QoL
Return to work | 12 months
  Rate of patients returning to work at 1 year (full time and / or medical part-time)
Body function - Pain intensity | 12 months
  Defined by International Classification of Functioning, Disability and Health (ICF), assessed by SF-BPI ; pain intensity (severity, means of 4 first items) and the impact of pain on functioning (interference, mean of the seven interference items on a 0-10 scale) ; higher scores mean higher pain (severity or interference)
Body function - CRPS severity score | 12 months
  Defined by Harden et al., signs + symptoms, 0 to 16 scale ; higher score means higher severity

CONTACTS AND LOCATIONS:
Overall Officials: Anne Berquin, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harden RN, Maihofner C, Abousaad E, Vatine JJ, Kirsling A, Perez RSGM, Kuroda M, Brunner F, Stanton-Hicks M, Marinus J, van Hilten JJ, Mackey S, Birklein F, Schlereth T, Mailis-Gagnon A, Graciosa J, Connoly SB, Dayanim D, Massey M, Frank H, Livshitz A, Bruehl S. A prospective, multisite, international validation of the Complex Regional Pain Syndrome Severity Score. Pain. 2017 Aug;158(8):1430-1436. doi: 10.1097/j.pain.0000000000000927. PMID 28715350
- [Background] Bean DJ, Johnson MH, Heiss-Dunlop W, Kydd RR. Extent of recovery in the first 12 months of complex regional pain syndrome type-1: A prospective study. Eur J Pain. 2016 Jul;20(6):884-94. doi: 10.1002/ejp.813. Epub 2015 Nov 2. PMID 26524108
- [Background] Brunner F, Bachmann LM, Perez RSGM, Marinus J, Wertli MM. Painful swelling after a noxious event and the development of complex regional pain syndrome 1: A one-year prospective study. Eur J Pain. 2017 Oct;21(9):1611-1617. doi: 10.1002/ejp.1064. Epub 2017 Jun 2. PMID 28573699
- [Background] Brunner F, Bachmann LM, Weber U, Kessels AG, Perez RS, Marinus J, Kissling R. Complex regional pain syndrome 1--the Swiss cohort study. BMC Musculoskelet Disord. 2008 Jun 23;9:92. doi: 10.1186/1471-2474-9-92. PMID 18573212
- [Background] Bruehl S, Maihofner C, Stanton-Hicks M, Perez RS, Vatine JJ, Brunner F, Birklein F, Schlereth T, Mackey S, Mailis-Gagnon A, Livshitz A, Harden RN. Complex regional pain syndrome: evidence for warm and cold subtypes in a large prospective clinical sample. Pain. 2016 Aug;157(8):1674-81. doi: 10.1097/j.pain.0000000000000569. PMID 27023422
- [Derived] Louis MH, Legrain V, Aron V, Filbrich L, Mouraux A, Henrard S, Guillaume L, Mouraux D, Barbier O, Libouton X, Berquin A. Complex regional pain syndrome evolution is determined by both biological and psychosocial factors: a 1-year prospective observational study. Pain. 2026 Feb 1;167(2):396-413. doi: 10.1097/j.pain.0000000000003815. Epub 2025 Oct 8. PMID 41065599